CLINICAL TRIAL: NCT04739319
Title: Project AMD: Comprehensive Characterisation of Age-Related Macular Degeneration and Its Progression
Acronym: Project AMD
Status: Recruiting | Type: Observational
Sponsor: Center for Eye Research Australia (Other)
Responsible Party: Sponsor
Other Study IDs: CenterERA
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Age Related Macular Degeneration; Geographic Atrophy; AMD; Age-related Macular Degeneration
Keywords: Age Related Macular Degeneration; Geographic Atrophy; Drusen; Macular disease
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, urine or tear samples will be obtained, on selected participants, to obtain genetic information and systematic markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age-Related Macular Degeneration: Participants with Age-Related Macular Degeneration
  Interventions: Other: N/A Observational study

INTERVENTIONS:
Other: N/A Observational study — N/A Observational study

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of irreversible vision loss worldwide, and nearly two million Australians have some signs of AMD. This proposed project is a prospective, observational study that seeks to to understand the underlying aetiology of AMD, factors associated with differences between age-related macular degeneration (AMD) phenotypes or severities, or between AMD and healthy individuals. It also seeks to understand the natural history of AMD progression and the factors associated with the rate of progression. In this project, the disease phenotype, genotype and severity and rate of progression will be determined based on non-invasive clinical imaging or functional assessment of the retina, from obtaining biological samples from the participants, or from patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older; and
2. either AMD (defined as having at least a medium druse >63 um), or having eyes with normal ageing changes (including small drusen ≤63 um) or no abnormalities as control participants

Exclusion Criteria:

1. ocular or systemic conditions other than AMD that could compromise retinal assessment or assessment of AMD and its progression; or
2. any participant with any mental or physical impairment that prevents them from signing an informed consent form or participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People in Australia aged 18 years or older with AMD or healthy controls, willing and able to provide informed consent, and willing to accept the study requirements.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2040-11 (Estimated); Study Completion 2040-11 (Estimated)

PRIMARY OUTCOMES:
Investigate the underlying aetiology of Age-Related Macular Degeneration | Up to 20 years
  The first aim of this project is to comprehensively investigate the underlying aetiology of AMD, characterise the AMD phenotype by understanding the differences between those with AMD and healthy individuals.
Characterise the natural history of Age-Related Macular Degeneration and factors associated with its rate of progression. | Up to 20 years
  The second aim of this project is to characterise the natural history of AMD and factors associated with its rate of progression. These aims will be achieved by using performing imaging and functional assessment of the retina, characterisation of the genetic, systemic and environmental factors, and by obtaining patient-reported outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Eye Research Australia, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD at the discretion of the Principal Investigator in a de-identified format

REFERENCES:
- See also: Related Info — https://www.cera.org.au/trials/project-amd-comprehensive-characterisation-of-age-related-macular-degeneration-and-its-progression/